CLINICAL TRIAL: NCT01648764
Title: Phase 1 Dose Escalation Study of LY2334737 Using 2 Dosing Regimens in Patients With Advanced and/or Metastatic Solid Tumors
Brief Title: A Study of LY2334737 in Participants With Cancer That is Advanced and/or Has Spread
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11967; 2008-000807-28 (EudraCT Number); I1C-MC-JLBE (Other: Eli Lilly & Company)
Record Dates: First submitted 2012-07-20; First posted 2012-07-24 (Estimated); Results first posted 2019-06-17 (Actual); Last update posted 2019-06-17 (Actual); Status verified 2019-03

CONDITIONS: Malignant Solid Tumor; Solid Tumor; Metastatic Tumor
MeSH Terms: conditions — Neoplasm Metastasis | interventions — LY2334737

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- LY2334737 - Arm A (Experimental): LY2334737 administered orally at escalating doses [40 milligrams (mg) - 200 mg] every other day for 21 days followed by 7 days without study drug (28 day treatment cycle). Participants may receive additional treatment cycles until discontinuation criterion is met.
  Interventions: Drug: LY2334737
- LY2334737 - Arm B (Experimental): LY2334737 administered orally at escalating doses (40 mg - 200 mg) every day for 7 days followed by 7 days without study drug then repeated (28 day treatment cycle). Participants may receive additional treatment cycles until discontinuation criterion is met.
  Interventions: Drug: LY2334737

INTERVENTIONS:
Drug: LY2334737 — Administered orally

SUMMARY:
The purpose of this study is to evaluate two different dosing regimens of LY2334737 in participants with cancer that is advanced and/or has spread to other parts of the body. Information about side effects will be collected.

DETAILED DESCRIPTION:
This study will consist of a Dose Escalation Phase (Arms A and B) followed by a Dose Confirmation Phase.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of advanced and/or metastatic cancer (including lymphoma) for which no treatment of higher priority exists
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2
* Estimated life expectancy of more than 12 weeks
* Have discontinued all previous therapies for cancer for at least 30 days (6 weeks for mitomycin-C or nitrosoureas) and recovered from acute effects of therapy
* Have discontinued radiotherapy more than one week before enrolling in the study and have recovered from the acute effects of therapy
* Have adequate organ function
* Follow your doctor's directions and live close enough to the study site so you can continue to go to the clinic for follow-up
* Are willing and able to swallow capsules and follow study procedures
* Have given written informed consent prior to any study-specific procedures
* Males and females with reproductive potential should use medically approved contraceptive precautions during the study and for 6 months following the last dose of study drug
* Females with child-bearing potential must have had a negative urine or serum pregnancy test 7 days prior to the first dose of study drug

Exclusion Criteria:

* Have gastrointestinal diseases or prior surgery that may interfere with the absorption of medication taken by mouth
* Females who are pregnant or lactating
* Symptomatic central nervous system malignancy or metastasis
* Known positive test results in human immunodeficiency virus (HIV), hepatitis B surface antigen (HBSAg), or hepatitis C antibodies (HCAb)
* Liver cirrhosis or chronic hepatitis
* Acute or chronic leukemia
* Are currently receiving treatment with valproic acid (VPA) and its derivatives, or if you have a history of intolerance to VPA
* Known hypersensitivity to gemcitabine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2008-09; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (4):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Philadelphia, Pennsylvania, United States
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Clichy, France
- Germany (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Berlin
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nuremberg

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participant Flow is reporting discontinuation from study drug. Completed participants were all those who completed Cycle 1.
Groups:
- 40 mg LY - Arm A Dose Escalation: 40 milligrams (mg) LY2334737 (LY) administered orally every other day for 21 days followed by 7 days without study drug (28-day treatment cycle). Participants could have received additional treatment cycles until discontinuation criterion was met.
- 50 mg LY - Arm A Dose Escalation: 50 mg LY2334737 administered orally every other day for 21 days followed by 7 days without study drug (28-day treatment cycle). Participants could have received additional treatment cycles until discontinuation criterion was met.
- 60 mg LY - Arm A Dose Escalation: 60 mg LY2334737 administered orally every other day for 21 days followed by 7 days without study drug (28-day treatment cycle). Participants could have received additional treatment cycles until discontinuation criterion was met.
- 70 mg LY - Arm A Dose Escalation: 70 mg LY2334737 administered orally every other day for 21 days followed by 7 days without study drug (28-day treatment cycle). Participants could have received additional treatment cycles until discontinuation criterion was met.
- 80 mg LY - Arm A Dose Escalation: 80 mg LY2334737 administered orally every other day for 21 days followed by 7 days without study drug (28-day treatment cycle). Participants could have received additional treatment cycles until discontinuation criterion was met.
- 90 mg LY - Arm A Dose Escalation; 90 mg LY - Arm A Dose Confirmation: 90 mg LY2334737 administered orally every other day for 21 days followed by 7 days without study drug (28-day treatment cycle). Participants could have received additional treatment cycles until discontinuation criterion was met.
- 100 mg LY - Arm A Dose Escalation: 100 mg LY2334737 administered orally every other day for 21 days followed by 7 days without study drug (28-day treatment cycle). Participants could have received additional treatment cycles until discontinuation criterion was met.
- 40 mg LY - Arm B Dose Escalation: 40 mg LY2334737 administered orally every day for 7 days followed by 7 days without study drug then repeated (28-day treatment cycle). Participants could have received additional treatment cycles until discontinuation criterion was met.
- 50 mg LY - Arm B Dose Escalation: 50 mg LY2334737 administered orally every day for 7 days followed by 7 days without study drug then repeated (28-day treatment cycle). Participants could have received additional treatment cycles until discontinuation criterion was met.
- 60 mg LY - Arm B Dose Escalation: 60 mg LY2334737 administered orally every day for 7 days followed by 7 days without study drug then repeated (28-day treatment cycle). Participants could have received additional treatment cycles until discontinuation criterion was met.
- 70 mg LY - Arm B Dose Escalation: 70 mg LY2334737 administered orally every day for 7 days followed by 7 days without study drug then repeated (28-day treatment cycle). Participants could have received additional treatment cycles until discontinuation criterion was met.
- 80 mg LY - Arm B Dose Escalation: 80 mg LY2334737 administered orally every day for 7 days followed by 7 days without study drug then repeated (28-day treatment cycle). Participants could have received additional treatment cycles until discontinuation criterion was met.
- 90 mg LY - Arm B Dose Escalation: 90 mg LY2334737 administered orally every day for 7 days followed by 7 days without study drug then repeated (28-day treatment cycle). Participants could have received additional treatment cycles until discontinuation criterion was met.
Period: Overall Study
Arm/Group | 40 mg LY - Arm A Dose Escalation | 50 mg LY - Arm A Dose Escalation | 60 mg LY - Arm A Dose Escalation | 70 mg LY - Arm A Dose Escalation | 80 mg LY - Arm A Dose Escalation | 90 mg LY - Arm A Dose Escalation | 100 mg LY - Arm A Dose Escalation | 40 mg LY - Arm B Dose Escalation | 50 mg LY - Arm B Dose Escalation | 60 mg LY - Arm B Dose Escalation | 70 mg LY - Arm B Dose Escalation | 80 mg LY - Arm B Dose Escalation | 90 mg LY - Arm B Dose Escalation | 90 mg LY - Arm A Dose Confirmation
Started | 3 | 3 | 3 | 3 | 3 | 5 | 9 | 3 | 3 | 7 | 3 | 9 | 7 | 12
Received at Least 1 Dose of Study Drug | 3 | 3 | 3 | 3 | 3 | 5 | 9 | 3 | 3 | 7 | 3 | 9 | 7 | 12
Completed | 3 | 2 | 3 | 3 | 3 | 3 | 4 | 3 | 3 | 4 | 3 | 4 | 3 | 9
Not Completed | 0 | 1 | 0 | 0 | 0 | 2 | 5 | 0 | 0 | 3 | 0 | 5 | 4 | 3
Not completed — Progressive Disease | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 2 | 0 | 1 | 2 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 3 | 1 | 1
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Investigator Decision | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All enrolled participants.
Groups:
- 70 mg LY - Arm A Dose Escalation: 70 mg LY2334737 administered orally every other day for 21 days followed by 7 days without study drug (28 -ay treatment cycle). Participants could have received additional treatment cycles until discontinuation criterion was met.
- 90 mg LY2334737 - Arm A Dose Confirmation: 90 mg LY2334737 administered orally every other day for 21 days followed by 7 days without study drug (28-day treatment cycle). Participants could have received additional treatment cycles until discontinuation criterion was met.
- Total: Total of all reporting groups
Arm/Group | 40 mg LY - Arm A Dose Escalation | 50 mg LY - Arm A Dose Escalation | 60 mg LY - Arm A Dose Escalation | 70 mg LY - Arm A Dose Escalation | 80 mg LY - Arm A Dose Escalation | 90 mg LY - Arm A Dose Escalation | 100 mg LY - Arm A Dose Escalation | 40 mg LY - Arm B Dose Escalation | 50 mg LY - Arm B Dose Escalation | 60 mg LY - Arm B Dose Escalation | 70 mg LY - Arm B Dose Escalation | 80 mg LY - Arm B Dose Escalation | 90 mg LY - Arm B Dose Escalation | 90 mg LY2334737 - Arm A Dose Confirmation | Total
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 5 | 9 | 3 | 3 | 7 | 3 | 9 | 7 | 12 | 73
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.7 (3.8) | 60.0 (20.3) | 56.3 (11.2) | 49.7 (17.2) | 49.7 (9.6) | 68.2 (6.2) | 54.4 (11.1) | 55.7 (7.2) | 65.0 (5.0) | 60.1 (9.3) | 52.7 (20.0) | 66.0 (4.6) | 61.9 (9.8) | 63.0 (6.4) | 59.9 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1 | 1 | 0 | 2 | 3 | 1 | 0 | 1 | 1 | 6 | 4 | 4 | 25
  Male | 2 | 3 | 2 | 2 | 3 | 3 | 6 | 2 | 3 | 6 | 2 | 3 | 3 | 8 | 48
Race [Count of Participants; unit: Participants]
  Caucasian | 3 | 2 | 1 | 3 | 3 | 5 | 8 | 3 | 2 | 7 | 2 | 9 | 7 | 11 | 66
  African | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 3
  West Asian | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Hispanic | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 3
Eastern Cooperative Oncology Group (ECOG) [Count of Participants; unit: Participants] — ECOG Performance Status: 0=asymptomatic, fully active, can carry on all predisease performance without restrictions; 1=symptomatic, fully ambulatory, but restricted in physically strenuous activity, able to perform light/sedentary tasks; 2=symptomatic, ambulatory, capable of all self-care but unable to carry out work activities, up and about more than 50% of waking hours and in bed less than 50% of day.
  Participants
    0 | 3 | 2 | 3 | 3 | 1 | 3 | 4 | 2 | 3 | 4 | 1 | 5 | 2 | 7 | 43
    1 | 0 | 1 | 0 | 0 | 2 | 2 | 5 | 1 | 0 | 3 | 2 | 3 | 5 | 5 | 29
    2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Disease Stage [Count of Participants; unit: Participants] — Stage III -the cancer has spread to nearby tissue or spread to far away lymph nodes. Stage IV -the cancer has spread to other organs of the body such as the other lung, brain or liver.
  Participants
    Stage III | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 3 | 6
    Stage IV | 3 | 3 | 2 | 3 | 3 | 4 | 9 | 3 | 3 | 6 | 3 | 9 | 7 | 9 | 67
Country of Enrollment [Count of Participants; unit: Participants]
  France | 3 | 3 | 3 | 2 | 1 | 2 | 5 | 2 | 3 | 4 | 2 | 4 | 1 | 6 | 41
  Germany | 0 | 0 | 0 | 1 | 2 | 3 | 3 | 1 | 0 | 2 | 0 | 4 | 3 | 2 | 21
  United States | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 1 | 3 | 4 | 11

OUTCOME MEASURES:

1. Primary Outcome: Recommended Dose for Phase 2 Studies
Description: Recommended Phase 2 dose was determined by maximum tolerated dose (MTD). The MTD was the highest dose level at which <2 out of 6 participants experienced a dose-limiting toxicity (DLT) in Cycle 1. DLT was an adverse event (AE) during Cycle 1 that was likely related to LY2334737 and fulfilled any of the following criteria: Common Terminology Criteria for Adverse Events (CTCAE) ≥Grade 3 nonhematological (except nausea/vomiting controlled with treatment); Grade 3 neutropenia with fever or any Grade 4 neutropenia with or without fever; Grade 3 thrombocytopenia with ≥Grade 2 bleeding or Grade 4 thrombocytopenia with or without bleeding; A recovery period longer than 14 days from last dose of LY2334737 to values allowing Cycle 2 to start; Other significant drug-related toxicity deemed by investigator to be dose limiting or that caused the participant to withdraw from the study. Pharmacokinetics and pharmacodynamics (PK/PD) were also taken into consideration for Phase 2 recommended dose.
Time Frame: Baseline up to 28 days postdose in Cycle 1 (28-day cycle)
Population: All participants who received at least 1 dose of study drug during dose escalation and dose confirmation treatment arms.
Measure: Number; unit: mg every other day for 21 days
Groups:
- LY2334737: LY2334737 was administered as 2 Arms A and B. Participants in treatment Arm A were administered LY2334737 orally in escalating doses of 40 to 100 milligrams (mg) of LY2334737 every other day for 21 days followed by 7 days without study drug. Participants in treatment Arm B were administered LY2334737 orally in escalating doses of 40 to 90 mg every day for 7 days followed by 7 days without study drug and then repeated. Both treatment cycles were 28 days.
Arm/Group | LY2334737
Number analyzed (Participants) | 73
mg every other day for 21 days | 90

2. Secondary Outcome: Pharmacokinetics: Area Under the Concentration-Time Curve (AUC) for LY2334737
Description: AUC over the dosing interval (AUC0-Ƭ) of LY2334737 for Arm A (single dose) is 0 to 48 hours postdose. AUC0-Ƭ of LY2334737 for Arm B (multiple doses) is 0 to 24 hours postdose and AUC time 0 to infinity (AUC0-∞) for LY2334737.
Time Frame: Cycle 1 Day 1 (C1 D1): 0.5, 1.5, 2, 3.5, 7 24 hours postdose; Cycle 1 Day 21 (C1 D21): predose, 0.5, 2, 3 to 4, 7, 24 hours postdose of 28-day cycle
Population: All participants who received at least 1 dose of study drug and had AUC0-Ƭ and AUC0-∞ values.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms*hours per milliliter (ng*h/mL)
Groups:
- 90 mg LY - Arm A Dose Escalation and Dose Confirmation: 90 mg LY2334737 administered orally every other day for 21 days followed by 7 days without study drug (28-day treatment cycle). Participants could have received additional treatment cycles until discontinuation criterion was met.
Arm/Group | 40 mg LY - Arm A Dose Escalation | 50 mg LY - Arm A Dose Escalation | 60 mg LY - Arm A Dose Escalation | 70 mg LY - Arm A Dose Escalation | 80 mg LY - Arm A Dose Escalation | 90 mg LY - Arm A Dose Escalation and Dose Confirmation | 100 mg LY - Arm A Dose Escalation | 40 mg LY - Arm B Dose Escalation | 50 mg LY - Arm B Dose Escalation | 60 mg LY - Arm B Dose Escalation | 70 mg LY - Arm B Dose Escalation | 80 mg LY - Arm B Dose Escalation | 90 mg LY - Arm B Dose Escalation
Number analyzed (Participants) | 3 | 2 | 3 | 3 | 3 | 14 | 8 | 3 | 3 | 7 | 2 | 7 | 7
nanograms*hours per milliliter (ng*h/mL)
  C1 D1 AUC0-Ƭ | 188 (4) | 315 (34) | 250 (45) | 225 (32) | 279 (33) | 469 (58) | 429 (14) | 133 (70) | 154 (14) | 312 (27) | 437 (89) | 232 (54) | 455 (35)
  C1 D1 AUC0-∞ | 188 (4) | 315 (34) | 250 (45) | 225 (32) | 279 (33) | 469 (58) | 429 (14) | 134 (71) | 156 (15) | 314 (27) | 440 (89) | 234 (54) | 460 (35)
  C1 D21, AUC0-Ƭ: number analyzed (Participants) | 3 | 2 | 3 | 2 | 3 | 13 | 3 | 3 | 3 | 5 | 2 | 5 | 3
  C1 D21, AUC0-Ƭ | 219 (31) | 364 (2) | 188 (76) | 318 (22) | 341 (76) | 525 (93) | 647 (47) | 227 (72) | 233 (12) | 445 (20) | 620 (119) | 392 (31) | 580 (31)

3. Secondary Outcome: Pharmacokinetics: Area Under the Concentration-Time Curve (AUC) for 2'2'-Difluorodeoxycytidine (dFdC)
Description: AUC over the dosing interval (AUC0-Ƭ) of dFdC (a metabolite of LY2334737) for Arm A (following a single dose of LY2334737) AUC0-Ƭ is 0-48 hours postdose, Arm B (following multiple doses of LY2334737) AUC 0-Ƭ is 0-24 hours postdose and AUC from time 0 to infinity (AUC0-∞).
Time Frame: Cycle 1 Day 1 (C1 D1): 0.5, 1.5, 2, 3.5, 7 24 hours post dose; Cycle 1 Day 21 (C1 D21): predose, 0.5, 2, 3 to 4, 7, 24 hours post dose of 28-day cycle
Population: All participants who received at least 1 dose of study drug and had AUC 0-Ƭ and AUC 0-∞ values.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms*hours/milliliter (ng*h/mL)
Arm/Group | 40 mg LY - Arm A Dose Escalation | 50 mg LY - Arm A Dose Escalation | 60 mg LY - Arm A Dose Escalation | 70 mg LY - Arm A Dose Escalation | 80 mg LY - Arm A Dose Escalation | 90 mg LY - Arm A Dose Escalation and Dose Confirmation | 100 mg LY - Arm A Dose Escalation | 40 mg LY - Arm B Dose Escalation | 50 mg LY - Arm B Dose Escalation | 60 mg LY - Arm B Dose Escalation | 70 mg LY - Arm B Dose Escalation | 80 mg LY - Arm B Dose Escalation | 90 mg LY - Arm B Dose Escalation
Number analyzed (Participants) | 3 | 2 | 3 | 3 | 3 | 14 | 7 | 3 | 3 | 7 | 2 | 7 | 7
nanograms*hours/milliliter (ng*h/mL)
  C1 D1 AUC 0-Ƭ: number analyzed (Participants) | 1 | 0 | 3 | 3 | 3 | 14 | 7 | 3 | 3 | 7 | 1 | 7 | 7
  C1 D1 AUC 0-Ƭ | 12.1 (NA) — Result is for 1 participant only. |  | 30.8 (54) | 30.7 (13) | 25.4 (45) | 54.9 (65) | 59.4 (14) | 21.2 (108) | 19.3 (25) | 27.2 (15) | 52.1 (NA) — Result is for 1 participant only. | 24.9 (46) | 46.0 (28)
  C1 D1 AUC 0-∞: number analyzed (Participants) | 1 | 0 | 3 | 3 | 3 | 14 | 7 | 3 | 3 | 7 | 1 | 7 | 7
  C1 D1 AUC 0-∞ | 12.1 (NA) — Results is for 1 participant only |  | 30.7 (54) | 30.7 (14) | 25.3 (46) | 54.8 (65) | 59.1 (15) | 21.1 (109) | 19.2 (24) | 27.2 (15) | 54.7 (NA) — Result is for 1 participant only. | 25.4 (46) | 46.4 (27)
  C1 D21 AUC 0-Ƭ: number analyzed (Participants) | 3 | 2 | 1 | 2 | 1 | 13 | 3 | 1 | 3 | 5 | 1 | 5 | 1
  C1 D21 AUC 0-Ƭ | 12.5 (30) | 26.6 (30) | 31.1 (NA) — Results is for 1 participant only. | 35.7 (18) | 53.4 (NA) — Results is for 1 participant only. | 59.6 (90) | 55.6 (67) | 38.6 (NA) — Results is for 1 participant only. | 27.8 (37) | 28.9 (8) | 74.8 (NA) — Results is for 1 participant only. | 45.5 (102) | 119 (NA) — Results is for 1 participant only.

4. Secondary Outcome: Pharmacokinetics: Area Under the Concentration-Time Curve (AUC) for Difluorodeoxyuridine (dFdU)
Description: Daily AUC from time 0 to 24 hours (AUC 0-24) of dFdU (a metabolite of LY2334737) for Arm A (single dose of LY2334737) and Arm B (multiple doses of LY2334737).
Time Frame: as for outcome 2
Population: All participants who received at least 1 dose of study drug and had AUC0-24 dFdU results.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms*hours per milliliter (ng*h/mL)
Groups:
- 40 mg LY - Arm A Dose Escalation: 40 milligram (mg) LY2334737 (LY) administered orally every other day for 21 days followed by 7 days without study drug (28-day treatment cycle). Participants could have received additional treatment cycles until discontinuation criterion was met.
Arm/Group | 40 mg LY - Arm A Dose Escalation | 50 mg LY - Arm A Dose Escalation | 60 mg LY - Arm A Dose Escalation | 70 mg LY - Arm A Dose Escalation | 80 mg LY - Arm A Dose Escalation | 90 mg LY - Arm A Dose Escalation and Dose Confirmation | 100 mg LY - Arm A Dose Escalation | 40 mg LY - Arm B Dose Escalation | 50 mg LY - Arm B Dose Escalation | 60 mg LY - Arm B Dose Escalation | 70 mg LY - Arm B Dose Escalation | 80 mg LY - Arm B Dose Escalation | 90 mg LY - Arm B Dose Escalation
Number analyzed (Participants) | 3 | 2 | 3 | 3 | 3 | 14 | 8 | 3 | 3 | 7 | 3 | 7 | 7
nanograms*hours per milliliter (ng*h/mL)
  C1 D1: number analyzed (Participants) | 3 | 2 | 3 | 3 | 3 | 14 | 8 | 3 | 3 | 7 | 2 | 7 | 7
  C1 D1 | 4990 (3) | 7250 (20) | 8060 (48) | 10800 (23) | 9350 (30) | 11500 (35) | 10800 (37) | 6080 (16) | 7020 (6) | 8660 (16) | 9620 (3) | 9370 (39) | 12400 (11)
  C1 D 21: number analyzed (Participants) | 3 | 2 | 3 | 2 | 3 | 13 | 3 | 3 | 3 | 5 | 2 | 5 | 3
  C1 D 21 | 22300 (31) | 21500 (49) | 24800 (18) | 26100 (4) | 21200 (57) | 28300 (38) | 29800 (23) | 29300 (37) | 32200 (2) | 35700 (37) | 37100 (27) | 35600 (27) | 39900 (35)

5. Secondary Outcome: Pharmacokinetics: Maximum Plasma Concentration (Cmax)
Description: Cmax for LY2334737 and its metabolites 2'2'-difluorodeoxycytidine (dFdC) and difluorodeoxyuridine (dFdU).
Time Frame: as for outcome 2
Population: All participants who received at least 1 dose of study drug and had Cmax values.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Arm/Group | 40 mg LY - Arm A Dose Escalation | 50 mg LY - Arm A Dose Escalation | 60 mg LY - Arm A Dose Escalation | 70 mg LY - Arm A Dose Escalation | 80 mg LY - Arm A Dose Escalation | 90 mg LY - Arm A Dose Escalation and Dose Confirmation | 100 mg LY - Arm A Dose Escalation | 40 mg LY - Arm B Dose Escalation | 50 mg LY - Arm B Dose Escalation | 60 mg LY - Arm B Dose Escalation | 70 mg LY - Arm B Dose Escalation | 80 mg LY - Arm B Dose Escalation | 90 mg LY - Arm B Dose Escalation
Number analyzed (Participants) | 3 | 2 | 3 | 3 | 3 | 14 | 8 | 3 | 3 | 7 | 2 | 7 | 7
nanogram per milliliter (ng/mL)
  C1 D1-LY2334737 | 53.9 (40) | 62.6 (79) | 72.4 (75) | 91.8 (96) | 118 (92) | 171 (105) | 89.3 (72) | 46.5 (33) | 79.4 (8) | 112 (37) | 134 (192) | 55.1 (51) | 163 (44)
  C1 D21-LY2334737: number analyzed (Participants) | 3 | 2 | 3 | 2 | 3 | 13 | 3 | 3 | 3 | 5 | 2 | 5 | 3
  C1 D21-LY2334737 | 68.4 (11) | 110 (41) | 35.7 (165) | 93.1 (43) | 61.5 (473) | 126 (71) | 147 (26) | 48.8 (102) | 37.9 (118) | 106 (42) | 108 (51) | 74.4 (46) | 137 (62)
  C1 D1-dFdC: number analyzed (Participants) | 3 | 2 | 3 | 3 | 3 | 14 | 7 | 3 | 3 | 7 | 2 | 7 | 7
  C1 D1-dFdC | 3.39 (35) | 4.83 (60) | 6.55 (109) | 13.0 (27) | 10.4 (72) | 16.0 (77) | 12.1 (91) | 10.9 (19) | 10.6 (26) | 11.2 (29) | 9.35 (69) | 6.14 (60) | 16.0 (43)
  C1 D21-dFdC: number analyzed (Participants) | 3 | 2 | 3 | 2 | 2 | 13 | 3 | 3 | 3 | 5 | 2 | 5 | 3
  C1 D21-dFdC | 3.64 (19) | 8.22 (4) | 3.94 (180) | 11.3 (33) | 10.9 (243) | 10.2 (80) | 10.9 (76) | 5.81 (131) | 4.05 (64) | 6.99 (39) | 7.03 (17) | 6.93 (46) | 16.7 (125)
  C1 D1-dFdU | 262 (6) | 393 (24) | 419 (42) | 532 (27) | 467 (23) | 594 (29) | 564 (27) | 305 (14) | 369 (13) | 442 (24) | 485 (10) | 466 (37) | 620 (11)
  C1 D21-dFdU: number analyzed (Participants) | 3 | 2 | 3 | 2 | 3 | 13 | 3 | 3 | 3 | 5 | 2 | 5 | 3
  C1 D21-dFdU | 1060 (25) | 992 (51) | 1120 (18) | 1330 (20) | 1050 (52) | 1390 (35) | 1360 (19) | 1450 (38) | 1670 (6) | 1650 (32) | 1690 (29) | 1680 (26) | 1940 (28)

6. Secondary Outcome: Number of Participants With Best Overall Response (BOR)
Description: Response defined using Response Evaluation Criteria in Solid Tumors (RECIST v1.0) criteria. Complete Response defined as disappearance of all target and non-target lesions and normalization of tumor marker level. Partial Response defined as ≥30% decrease in sum of the longest diameter (LD) of target lesions, taking as reference the baseline sum LD. Progressive Disease (PD) defined as ≥20% increase in the sum of the LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of 1 or more new lesions, or appearance of 1 or more new lesions and/or unequivocal progression of existing non-target lesions. Stable Disease was defined as small changes that did not meet above criteria and unknown defined as response status was not known. The BOR was the best response recorded from the start of the treatment until disease progression/recurrence (taking as reference for PD the smallest measurements recorded since the treatment started).
Time Frame: Baseline to measured disease progression up to 33 weeks
Population: All participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | 40 mg LY - Arm A Dose Escalation | 50 mg LY - Arm A Dose Escalation | 60 mg LY - Arm A Dose Escalation | 70 mg LY - Arm A Dose Escalation | 80 mg LY - Arm A Dose Escalation | 90 mg LY - Arm A Dose Escalation | 100 mg LY - Arm A Dose Escalation | 40 mg LY - Arm B Dose Escalation | 50 mg LY - Arm B Dose Escalation | 60 mg LY - Arm B Dose Escalation | 70 mg LY - Arm B Dose Escalation | 80 mg LY - Arm B Dose Escalation | 90 mg LY - Arm B Dose Escalation | 90 mg LY - Arm A Dose Confirmation
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 5 | 9 | 3 | 3 | 7 | 3 | 9 | 7 | 12
Participants
  Complete Response | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Partial Response | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Stable Disease | 1 | 2 | 2 | 0 | 1 | 0 | 1 | 0 | 1 | 2 | 1 | 0 | 0 | 0
  Progressive Disease | 2 | 1 | 1 | 3 | 2 | 2 | 4 | 3 | 2 | 3 | 2 | 3 | 4 | 10
  Unknown | 0 | 0 | 0 | 0 | 0 | 3 | 4 | 0 | 0 | 2 | 0 | 6 | 3 | 2

7. Secondary Outcome: Progression-Free Survival (PFS)
Description: PFS was defined as the time from date of first dose to the first observation of disease progression or death due to any cause.
  Due to the different tumor types, schedules and doses, the PFS was not analyzed.
Time Frame: Baseline to measured disease progression or death up to 33 weeks
Population: Zero participants analyzed. No data collected for PFS.
Arm/Group | 40 mg LY - Arm A Dose Escalation | 50 mg LY - Arm A Dose Escalation | 60 mg LY - Arm A Dose Escalation | 70 mg LY - Arm A Dose Escalation | 80 mg LY - Arm A Dose Escalation | 90 mg LY - Arm A Dose Escalation | 100 mg LY - Arm A Dose Escalation | 40 mg LY - Arm B Dose Escalation | 50 mg LY - Arm B Dose Escalation | 60 mg LY - Arm B Dose Escalation | 70 mg LY - Arm B Dose Escalation | 80 mg LY - Arm B Dose Escalation | 90 mg LY - Arm B Dose Escalation | 90 mg LY - Arm A Dose Confirmation
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

8. Secondary Outcome: Percentage of Participants With Changes in QT Interval (>30 Milliseconds) From Baseline
Description: Fridericia-corrected QT (QTcF) interval corrected for heart rate was assessed using triplicate 12-lead electrocardiograms (ECGs). Change in QT interval from baseline was calculated using a time matched approach, that is change from baseline was calculated by subtracting the respective reading taken at the same nominal time on Day-1 from the reading taken on Days 1 and 21; change from baseline was calculated by subtracting the last non-missing ECG assessment on or prior to Day 1, 0.5 hours prior to dose from assessment on Day 2 and Day 22. The outlying QTcF intervals were defined using the criteria: change from baseline in mean QTcF interval >30 milliseconds
Time Frame: Day -1: 24.5 hours, 22 hours and 17 hours predose; Cycle 1 Days 1 and 21, 0.5 hours predose, 2 hours, 7 hours and 24 hours postdose (28-day cycles)
Population: All participants who received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | 40 mg LY - Arm A Dose Escalation | 50 mg LY - Arm A Dose Escalation | 60 mg LY - Arm A Dose Escalation | 70 mg LY - Arm A Dose Escalation | 80 mg LY - Arm A Dose Escalation | 90 mg LY - Arm A Dose Escalation | 100 mg LY - Arm A Dose Escalation | 40 mg LY - Arm B Dose Escalation | 50 mg LY - Arm B Dose Escalation | 60 mg LY - Arm B Dose Escalation | 70 mg LY - Arm B Dose Escalation | 80 mg LY - Arm B Dose Escalation | 90 mg LY - Arm B Dose Escalation | 90 mg LY - Arm A Dose Confirmation
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 5 | 9 | 3 | 3 | 7 | 3 | 9 | 7 | 12
percentage of participants | 33.3 | 33.3 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 11.1 | 0.0 | 0.0

9. Other Pre Specified Outcome: Number of Participants With Dose-Limiting Toxicity (DLT)
Description: DLT was defined as an adverse event (AE) during Cycle 1 that was likely related to the LY2334737 and fulfilled any of the following criteria: Common Terminology Criteria for Adverse Events (CTCAE) ≥Grade 3 nonhematological (except nausea/vomiting controlled with treatment); Grade 3 neutropenia with fever or any Grade 4 neutropenia with or without fever; Grade 3 thrombocytopenia with ≥ Grade 2 bleeding or Grade 4 thrombocytopenia; with or without bleeding A recovery period longer than 14 days from the last dose of LY2334737 to values allowing Cycle 2 to start; other significant drug-related toxicity deemed by the investigator to be dose limiting or that caused the participant to withdraw from the study.
Time Frame: Cycle 1 (28-day cycle)
Population: All participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | 40 mg LY - Arm A Dose Escalation | 50 mg LY - Arm A Dose Escalation | 60 mg LY - Arm A Dose Escalation | 70 mg LY - Arm A Dose Escalation | 80 mg LY - Arm A Dose Escalation | 90 mg LY - Arm A Dose Escalation | 100 mg LY - Arm A Dose Escalation | 40 mg LY - Arm B Dose Escalation | 50 mg LY - Arm B Dose Escalation | 60 mg LY - Arm B Dose Escalation | 70 mg LY - Arm B Dose Escalation | 80 mg LY - Arm B Dose Escalation | 90 mg LY - Arm B Dose Escalation | 90 mg LY - Arm A Dose Confirmation
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 5 | 9 | 3 | 3 | 7 | 3 | 9 | 7 | 12
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 1 | 0 | 1 | 2 | 1

10. Secondary Outcome: Percentage of Participants With Changes in R-R Interval From Baseline
Description: Changes in R-R interval from baseline was calculated using a time matched approach, that is change from baseline was calculated by subtracting the respective reading taken at the same nominal time on Day -1 from the reading taken on Days 1 and 21; change from baseline was calculated by subtracting the last non-missing electrocardiogram (ECG) assessment on or prior to Day 1 and 0.5 hours prior to dose for Day 2 and Day 22. Percentage of participants with changes in R-R interval from baseline was calculated as the number of participants with a change not equal to 0 across all time points divided by the number of treated participants multiplied by 100.
Time Frame: Day -1: 24.5 hours, 22 hours and 17 hours predose; Cycle 1 Days 1 and 21: 0.5 hours predose, 2 hours, 7 hours and 24 hours postdose
Population: All participants who received at least 1 dose of study drug with R-R interval data at all time points.
Measure: Number; unit: percentage of participants
Groups:
- 90 mg LY - Arm A Dose Confirmation: 90 mg LY2334737 administered orally every day for 7 days followed by 7 days without study drug (28-day treatment cycle). Participants could have received additional treatment cycles until discontinuation criterion was met.
Arm/Group | 40 mg LY - Arm A Dose Escalation | 50 mg LY - Arm A Dose Escalation | 60 mg LY - Arm A Dose Escalation | 70 mg LY - Arm A Dose Escalation | 80 mg LY - Arm A Dose Escalation | 90 mg LY - Arm A Dose Escalation | 100 mg LY - Arm A Dose Escalation | 40 mg LY - Arm B Dose Escalation | 50 mg LY - Arm B Dose Escalation | 60 mg LY - Arm B Dose Escalation | 70 mg LY - Arm B Dose Escalation | 80 mg LY - Arm B Dose Escalation | 90 mg LY - Arm B Dose Escalation | 90 mg LY - Arm A Dose Confirmation
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 5 | 9 | 3 | 3 | 7 | 3 | 9 | 7 | 12
percentage of participants | 100.0 | 100.0 | 100.0 | 100.0 | 100.0 | 100.0 | 100.0 | 100.0 | 100.0 | 100.0 | 100.0 | 100.0 | 100.0 | 100.0

11. Secondary Outcome: Pharmacokinetics: Minimum Plasma Concentration (Cmin)
Description: Cmin for LY2334737 and its metabolite 2'2'-difluorodeoxycytidine (dFdC).
Time Frame: Cycle 1 Day 1 (C1 D1): 0.5, 1.5, 2, 3.5, 7, 24 hours postdose; Cycle 1 Day 21 (C1 D21): predose, 0.5, 2, 3 to 4, 7, 24 hours postdose of 28-day cycle
Population: All participants who received at least 1 dose of study drug and had Cmin values
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per milliliter (ng/mL)
Arm/Group | 40 mg LY - Arm A Dose Escalation | 50 mg LY - Arm A Dose Escalation | 60 mg LY - Arm A Dose Escalation | 70 mg LY - Arm A Dose Escalation | 80 mg LY - Arm A Dose Escalation | 90 mg LY - Arm A Dose Escalation and Dose Confirmation | 100 mg LY - Arm A Dose Escalation | 40 mg LY - Arm B Dose Escalation | 50 mg LY - Arm B Dose Escalation | 60 mg LY - Arm B Dose Escalation | 70 mg LY - Arm B Dose Escalation | 80 mg LY - Arm B Dose Escalation | 90 mg LY - Arm B Dose Escalation
Number analyzed (Participants) | 3 | 2 | 3 | 3 | 3 | 14 | 8 | 3 | 3 | 7 | 2 | 7 | 7
nanograms per milliliter (ng/mL)
  C1 D1 LY | 0.451 (129) | 0.319 (10) | 0.458 (43) | 0.279 (66) | 0.392 (15) | 0.901 (94) | 0.920 (45) | 0.379 (118) | 0.279 (98) | 0.456 (36) | 0.773 (57) | 0.665 (80) | 0.898 (84)
  C1 D21 LY: number analyzed (Participants) | 3 | 2 | 3 | 2 | 3 | 13 | 3 | 3 | 3 | 5 | 2 | 5 | 3
  C1 D21 LY | 0.264 (34) | 0.223 (89) | 0.519 (1479) | 1.01 (59) | 0.568 (18) | 1.04 (146) | 0.934 (274) | 0.347 (148) | 0.523 (43) | 1.50 (66) | 0.347 (251) | 1.04 (89) | 0.561 (395)
  C1 D1 dFdC: number analyzed (Participants) | 3 | 2 | 3 | 3 | 3 | 14 | 7 | 3 | 3 | 7 | 2 | 7 | 7
  C1 D1 dFdC | 0.774 (52) | 1.89 (28) | 0.507 (47) | 0.891 (45) | 0.918 (56) | 0.901 (108) | 0.928 (179) | 1.45 (49) | 0.567 (53) | 1.10 (60) | 0.840 (133) | 0.809 (99) | 1.65 (134)
  C1 D21 dFdC: number analyzed (Participants) | 3 | 2 | 3 | 2 | 2 | 13 | 3 | 3 | 3 | 5 | 2 | 5 | 3
  C1 D21 dFdC | 0.431 (24) | 0.949 (47) | 1.25 (37) | 0.612 (198) | 1.87 (155) | 0.647 (107) | 0.643 (76) | 1.21 (170) | 0.409 (82) | 1.19 (112) | 0.804 (363) | 1.49 (80) | 2.96 (180)

ADVERSE EVENTS:
Description: Study-specific clinical outcomes due to progressive disease were not considered to be a serious adverse event (SAE) unless the investigator deemed it related to the use of the study drug.
Groups:
- 40 mg LY - Arm A Dose Escalation: 40 milligrams (mg) LY2334737 administered orally every other day for 21 days followed by 7 days without study drug (28-day treatment cycle). Participants could have received additional treatment cycles until discontinuation criterion was met.
Arm/Group | 40 mg LY - Arm A Dose Escalation | 50 mg LY - Arm A Dose Escalation | 60 mg LY - Arm A Dose Escalation | 70 mg LY - Arm A Dose Escalation | 80 mg LY - Arm A Dose Escalation | 90 mg LY - Arm A Dose Escalation | 100 mg LY - Arm A Dose Escalation | 40 mg LY - Arm B Dose Escalation | 50 mg LY - Arm B Dose Escalation | 60 mg LY - Arm B Dose Escalation | 70 mg LY - Arm B Dose Escalation | 80 mg LY - Arm B Dose Escalation | 90 mg LY - Arm B Dose Escalation | 90 mg LY - Arm A Dose Confirmation
Serious Adverse Events (participants affected / at risk) | 2/3 | 1/3 | 1/3 | 1/3 | 1/3 | 5/5 | 5/9 | 1/3 | 1/3 | 2/7 | 2/3 | 5/9 | 6/7 | 6/12
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 3/3 | 3/3 | 3/3 | 5/5 | 9/9 | 3/3 | 3/3 | 7/7 | 3/3 | 9/9 | 6/7 | 12/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 40 mg LY - Arm A Dose Escalation (N=3) | 50 mg LY - Arm A Dose Escalation (N=3) | 60 mg LY - Arm A Dose Escalation (N=3) | 70 mg LY - Arm A Dose Escalation (N=3) | 80 mg LY - Arm A Dose Escalation (N=3) | 90 mg LY - Arm A Dose Escalation (N=5) | 100 mg LY - Arm A Dose Escalation (N=9) | 40 mg LY - Arm B Dose Escalation (N=3) | 50 mg LY - Arm B Dose Escalation (N=3) | 60 mg LY - Arm B Dose Escalation (N=7) | 70 mg LY - Arm B Dose Escalation (N=3) | 80 mg LY - Arm B Dose Escalation (N=9) | 90 mg LY - Arm B Dose Escalation (N=7) | 90 mg LY - Arm A Dose Confirmation (N=12)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Colonic obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Gastric haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Proctocolitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Asthenia (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Disease progression (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
General physical health deterioration (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mucosal inflammation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Bile duct stenosis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cholangitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cholestasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cytokine release syndrome (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Klebsiella bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Electrocardiogram qt prolonged (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Troponin t increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Exeresis (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 40 mg LY - Arm A Dose Escalation (N=3) | 50 mg LY - Arm A Dose Escalation (N=3) | 60 mg LY - Arm A Dose Escalation (N=3) | 70 mg LY - Arm A Dose Escalation (N=3) | 80 mg LY - Arm A Dose Escalation (N=3) | 90 mg LY - Arm A Dose Escalation (N=5) | 100 mg LY - Arm A Dose Escalation (N=9) | 40 mg LY - Arm B Dose Escalation (N=3) | 50 mg LY - Arm B Dose Escalation (N=3) | 60 mg LY - Arm B Dose Escalation (N=7) | 70 mg LY - Arm B Dose Escalation (N=3) | 80 mg LY - Arm B Dose Escalation (N=9) | 90 mg LY - Arm B Dose Escalation (N=7) | 90 mg LY - Arm A Dose Confirmation (N=12)
Anaemia (Blood and lymphatic system disorders) | 3 (4) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 3 (3) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 2 (3) | 3 (4) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (4) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hearing impaired (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Conjunctivitis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eyelid oedema (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 3 (3) | 1 (1) | 4 (4) | 1 (1) | 1 (1)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 3 (3) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 3 (3) | 1 (1) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 3 (3) | 2 (3) | 0 (0) | 2 (2) | 0 (0) | 3 (3) | 2 (2) | 3 (3)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal disorder (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Melaena (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (3) | 2 (3) | 1 (1) | 2 (2) | 2 (2) | 4 (4) | 7 (8) | 1 (1) | 1 (1) | 2 (2) | 2 (5) | 3 (3) | 4 (4) | 6 (6)
Obstruction gastric (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral disorder (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis chronic (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Subileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (3) | 2 (2) | 0 (0) | 1 (4) | 2 (2) | 5 (5) | 6 (7) | 2 (2) | 1 (1) | 1 (1) | 2 (3) | 4 (4) | 2 (2) | 3 (3)
Asthenia (General disorders) | 2 (3) | 2 (2) | 3 (4) | 2 (2) | 1 (1) | 2 (2) | 4 (4) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 4 (4) | 1 (1) | 4 (4)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chills (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (2) | 0 (0) | 2 (2) | 1 (1) | 3 (3) | 1 (1) | 3 (3)
Condition aggravated (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Face oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 3 (3) | 4 (4) | 1 (1) | 0 (0) | 1 (2) | 1 (1) | 2 (2) | 1 (1) | 3 (3)
General physical health deterioration (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 3 (3)
Mucosal inflammation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Multi-organ failure (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oedema (General disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 3 (5) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 2 (2) | 1 (2) | 2 (2)
Pyrexia (General disorders) | 2 (4) | 2 (2) | 2 (2) | 3 (6) | 1 (2) | 1 (1) | 2 (2) | 2 (4) | 3 (4) | 4 (5) | 2 (2) | 4 (5) | 3 (3) | 6 (6)
Cholestasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Jaundice (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fungal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Genital herpes (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Herpes virus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral herpes (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Staphylococcal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Activated partial thromboplastin time prolonged (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 3 (4) | 2 (2) | 1 (1) | 0 (0) | 2 (3) | 0 (0) | 2 (2) | 3 (3) | 1 (1) | 2 (2) | 1 (1) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 2 (3) | 2 (2) | 0 (0) | 1 (1) | 3 (4) | 1 (1) | 2 (2) | 3 (3) | 1 (1) | 3 (3) | 1 (1) | 0 (0)
Blood albumin decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 2 (3) | 1 (1) | 0 (0) | 3 (3) | 1 (1) | 2 (2) | 2 (2) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood calcium decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Blood magnesium decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Blood phosphorus decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood potassium decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood sodium decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
C-reactive protein increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Eastern cooperative oncology group performance status worsened (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Haemoglobin decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
International normalised ratio increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neutrophil count increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Prothrombin time prolonged (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 3 (3) | 0 (0) | 2 (2)
Decreased appetite (Metabolism and nutrition disorders) | 2 (2) | 3 (3) | 2 (2) | 1 (2) | 2 (2) | 3 (4) | 3 (3) | 1 (1) | 1 (1) | 4 (4) | 1 (1) | 7 (7) | 1 (1) | 3 (3)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperuricaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 3 (4) | 3 (3) | 3 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (4) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 2 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malnutrition (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ataxia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Balance disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Convulsion (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Extrapyramidal disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 1 (1)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Speech disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 1 (1) | 0 (0)
Bladder obstruction (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Proteinuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 4 (4)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hot flush (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Jugular vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral coldness (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Phlebitis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days